CLINICAL TRIAL: NCT01056510
Title: A Randomized Study to Assess the Effect on Response Rate of MabThera (Rituximab) Added to a Standard Chemotherapy, Bendamustine or Chlorambucil, in Patients With Chronic Lymphocytic Leukemia
Brief Title: A Study of MabThera Added to Bendamustine or Chlorambucil in Patients With Chronic Lymphocytic Leukemia (MaBLe)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO22468; 2009-012072-28
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Chlorambucil; Rituximab

ARMS (2):
- A (Experimental)
  Interventions: Drug: bendamustine; Drug: rituximab [MabThera/Rituxan]
- B (Experimental)
  Interventions: Drug: chlorambucil; Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: bendamustine — 90mg/m2 (first-line) or 70mg/m2 (second-line) iv, days 1 and 2 every 4 weeks, cycles 1-6
  Arms: A
Drug: chlorambucil — 10mg/m2 po days 1-7 every 4 weeks, for up to 12 cycles
  Arms: B
Drug: rituximab [MabThera/Rituxan] — 375mg/m2 iv day 1 of cycle 1, followed by 500mg/m2 iv every 4 weeks cycles 2-6

SUMMARY:
This randomized, open-label, parallel group study will assess the effect on response rate and the safety of MabThera added to either bendamustine or chlorambucil in patients with chronic lymphocytic leukemia. Patients will be randomized to receive six 4-week cycles of either A) MabThera (375mg/m2 iv day 1 of cycle 1, 500mg/m2 iv cycles 2-6) plus bendamustine (90mg/m2 as first-line or 70mg/m2 as second-line therapy, iv on days 1 and 2, cycles 1-6), or B)MabThera plus chlorambucil (10mg/m2 po daily, days 1-7, cycles 1-6). Patients in group B can receive up to 6 further cycles of chlorambucil as monotherapy. Anticipated time on study treatment is 6-12 months, and target sample size is 600-700 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=18 years of age
* chronic lymphocytic leukemia
* active CLL with progressive Binet stage B or C
* ineligible for treatment with fludarabine
* for second line patients, only pretreatment with rituximab and/or chlorambucil is allowed
* EOCG performance status >/=2

Exclusion Criteria:

* patients who have relapsed within <12 months of first dose of prior rituximab or chlorambucil first-line therapy
* previous or planned stem cell transplantation
* radioimmunotherapy within 6 months prior to starting study treatment
* transformation to aggressive B-cell malignancy
* any other concurrent anti-cancer therapy, or glucocorticoid >/=20mg daily prednisolone or equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (69):
- Finland (2):
  - Pori
  - Vantaa
- France (19):
  - Argenteuil
  - Avignon
  - Blois
  - Bordeaux
  - Brest
  - La Roche-sur-Yon
  - La Tronche
  - Le Mans
  - Lens
  - Limoges
  - Lyon
  - Marseille
  - Mulhouse
  - Nice
  - Nîmes
  - Paris
  - Perpignan
  - Pierre-Bénite
  - Salouël
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Spain (18):
  - Vitoria-Gasteiz, Alava
  - Elche, Alicante
  - Barcelona, Barcelona
  - Jerez de la Frontera, Cadiz
  - Torrelavega, Cantabria
  - Huelva, Huelva
  - A Coruña, La Coruña
  - León, Leon
  - Alcorcón, Madrid
  - Madrid, Madrid
  - Málaga, Malaga
  - Cartagena, Murcia
  - Murcia, Murcia
  - Salamanca, Salamanca
  - Seville, Sevilla
  - Tarragona, Tarragona
  - Valencia, Valencia
  - Zaragoza, Zaragoza
- Sweden (7):
  - Falun
  - Kristianstad
  - Luleå
  - Sundsvall
  - Uddevalla
  - Umeå
  - Uppsala
- Tunis, Tunisia
- Turkey (Türkiye) (8):
  - Ankara
  - Bursa
  - Edirne
  - Istanbul
  - Izmir
  - Kayseri
  - Kocaeli
  - Samsun
- United Kingdom (11):
  - Blackpool
  - Bournemouth
  - Edinburgh
  - Leeds
  - London
  - Maidstone
  - Manchester
  - Oxford
  - Romford
  - Somerset
  - Truro

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening examination was performed within 28 days before randomization. Participants who fulfilled all the inclusion and none of the exclusion criteria were randomized to one of the two treatment groups.
Groups:
- Rituximab + Bendamustine: Participants received a specialized first-line or second-line regimen based upon prior chemotherapy exposure. Participants received intravenous (IV) rituximab 375 milligrams per square meter (mg/m^2) on Day 1 of Cycle 1 and 500 mg/m^2 on Day 1 of Cycles 2 to 6. In those requiring a first-line regimen, bendamustine was administered IV at a dose of 90 mg/m^2 on Days 1 and 2 of Cycles 1 to 6. In those requiring a second-line regimen, the bendamustine dose was lowered to 70 mg/m^2. Each cycle was 4 weeks in duration. Treatment was discontinued early in participants who experienced progressive disease (PD).
- Rituximab + Chlorambucil: Participants received IV rituximab 375 mg/m^2 on Day 1 of Cycle 1 and 500 mg/m^2 on Day 1 of Cycles 2 to 6. Chlorambucil was administered orally (PO) at a dose of 10 mg/m^2 on Days 1 to 7, beginning with Cycle 1 and continuing for up to 12 cycles or until complete response (CR) was achieved. Each cycle was 4 weeks in duration. Treatment was discontinued early in participants who experienced PD.
Period: Overall Study
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Started | 178 | 179
Completed | 124 | 115
Not Completed | 54 | 64
Not completed — Dropout Before Start of Treatment | 1 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Death | 29 | 34
Not completed — Noncompliance | 1 | 3
Not completed — Physician Decision | 4 | 5
Not completed — Lost to Follow-up | 5 | 6
Not completed — Other | 10 | 12
Not completed — Missing | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: all randomized participants
Groups:
- Rituximab + Bendamustine: Participants received a specialized first-line or second-line regimen based upon prior chemotherapy exposure. Participants received IV rituximab 375 mg/m^2 on Day 1 of Cycle 1 and 500 mg/m^2 on Day 1 of Cycles 2 to 6. In those requiring a first-line regimen, bendamustine was administered IV at a dose of 90 mg/m^2 on Days 1 and 2 of Cycles 1 to 6. In those requiring a second-line regimen, the bendamustine dose was lowered to 70 mg/m^2. Each cycle was 4 weeks in duration. Treatment was discontinued early in participants who experienced PD.
- Rituximab + Chlorambucil: Participants received IV rituximab 375 mg/m^2 on Day 1 of Cycle 1 and 500 mg/m^2 on Day 1 of Cycles 2 to 6. Chlorambucil was administered PO at a dose of 10 mg/m^2 on Days 1 to 7, beginning with Cycle 1 and continuing for up to 12 cycles or until CR was achieved. Each cycle was 4 weeks in duration. Treatment was discontinued early in participants who experienced PD.
- Total: Total of all reporting groups
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil | Total
Number analyzed (Participants) | 178 | 179 | 357
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (9.87) | 70.1 (9.88) | 70.3 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 61 | 134
  Male | 105 | 118 | 223

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Confirmed Complete Response (CR) According to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 Guidelines in the First-Line Subpopulation After 6 Cycles of Therapy
Description: The definition of confirmed CR required all of the following criteria as assessed at least 2 months after completion of therapy: peripheral blood lymphocytes less than (<) 4 times 10^9 cells per liter (cells/L); absence of significant lymphadenopathy, hepatomegaly, or splenomegaly due to chronic lymphocytic leukemia (CLL) involvement; absence of constitutional symptoms; normal complete blood count (CBC) without need for transfusion or exogenous growth factors, as exhibited by neutrophils at least (>/=) 1.5 times 10^9 cells/L, platelets greater than (>) 100 times 10^9 cells/L, and hemoglobin > 11.0 grams per deciliter (g/dL); normocellular bone marrow (BM) aspirate with < 30 percent (%) lymphocytes; absence of lymphoid nodules; and BM biopsy without CLL activity. The percentage of participants achieving confirmed CR was calculated as the number of participants meeting the above criteria divided by the number of participants analyzed, multiplied by 100.
Time Frame: At least 2 months after completion of therapy (up to 32 weeks)
Population: ITT Population (First-Line Subpopulation): A subset of participants requiring a first-line regimen for CLL.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 121 | 120
percentage of participants
  Confirmed CR with biopsy | 24 | 9.2
  CR without biopsy | 2.5 | 5.8
  No confirmed CR | 73.6 | 85
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; The first-line subpopulation became the focus of the primary statistical analysis following the protocol amendment dated 21-May-2012; Test type: Superiority or Other; p = 0.002, Chi-squared, Corrected — Based on one-sided continuity corrected Chi-Square Test for participants achieving CR confirmed with biopsy versus those not achieving CR confirmed with biopsy

2. Secondary Outcome: Percentage of Participants Achieving Confirmed CR According to IWCLL 2008 Guidelines in the Pooled Population After 6 Cycles of Therapy
Description: The definition of confirmed CR required all of the following criteria as assessed at least 2 months after completion of therapy: peripheral blood lymphocytes < 4 times 10^9 cells/L; absence of significant lymphadenopathy, hepatomegaly, or splenomegaly due to CLL involvement; absence of constitutional symptoms; normal CBC without need for transfusion or exogenous growth factors, as exhibited by neutrophils >/= 1.5 times 10^9 cells/L, platelets > 100 times 10^9 cells/L, and hemoglobin > 11.0 g/dL; normocellular BM aspirate with < 30% lymphocytes; absence of lymphoid nodules; and BM biopsy without CLL activity. The percentage of participants achieving confirmed CR was calculated as the number of participants meeting the above criteria divided by the number of participants analyzed, multiplied by 100.
Time Frame: At least 2 months after completion of therapy (up to 32 weeks)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 178 | 179
percentage of participants
  Confirmed CR with biopsy | 21.3 | 6.7
  CR without biopsy | 2.8 | 4.5
  No confirmed CR | 75.8 | 88.8
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Achieving Confirmed CR According to IWCLL 2008 Guidelines in the Second-Line Subpopulation After 6 Cycles of Therapy
Description: as for outcome 2
Time Frame: At least 2 months after completion of therapy (up to 32 weeks)
Population: ITT Population (Second-Line Subpopulation): A subset of participants requiring a second-line regimen for CLL.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 57 | 59
percentage of participants
  Confirmed CR with biopsy | 15.8 | 1.7
  CR without biopsy | 3.5 | 1.7
  No confirmed CR | 80.7 | 96.6
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; Test type: Superiority or Other; p = 0.009, Chi-squared, Corrected — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants Achieving a Best Overall Response of CR, CR With Incomplete Marrow Recovery (CRi), Partial Response (PR), or Nodular PR (nPR) in the First-Line Subpopulation
Description: The criteria for CR are identified in previous outcome measure(s). Those fulfilling CR criteria but who have persistent anemia, thrombocytopenia, or neutropenia were considered CRi. The definition of PR required that the following be documented for minimum 2 months: >/= 50% decrease in peripheral blood lymphocytes from Baseline; reduction in lymphadenopathy; >/= 50% reduction in spleen or liver enlargement; and CBC with one of the following without need for transfusion or exogenous growth factors: polymorphonuclear leukocytes >/= 1.5 times 10^9 cells/L, platelets > 100 times 10^9 cells/L or >/= 50% improvement from Baseline, or hemoglobin > 11.0 g/dL or >/= 50% improvement from Baseline. Participants with lymphoid nodules who otherwise met CR criteria were considered nPR. The percentage of participants achieving each level of response was calculated as the number of participants meeting the above criteria divided by the number of participants analyzed, multiplied by 100.
Time Frame: After 3 and 6 treatment cycles and from Baseline to the end-of-treatment (EOT) visit, completed within 10 days before cutoff for data collection
Population: ITT Population (First-Line Subpopulation)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 121 | 120
percentage of participants
  After 3 cycles | 78.5 [70.1 to 85.5] | 80.0 [71.7 to 86.7]
  After 6 cycles | 75.2 [66.5 to 82.6] | 79.2 [70.8 to 86.0]
  At the EOT visit | 90.9 [84.3 to 95.4] | 85.8 [78.3 to 91.5]
Statistical Analysis 1: Comparison: Rituximab + Bendamustine; After 3 cycles; Test type: Superiority or Other; p = 0.900, Chi-squared, Corrected — Based on two-sided continuity corrected Chi-Square Test
Statistical Analysis 2: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; After 6 cycles; Test type: Superiority or Other; p = 0.563, Chi-squared, Corrected — Based on two-sided continuity corrected Chi-Square Test
Statistical Analysis 3: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; At the EOT visit; Test type: Superiority or Other; p = 0.304, Chi-squared, Corrected — Based on two-sided continuity corrected Chi-Square Test

5. Secondary Outcome: Percentage of Participants by Disease Response Category in the First-Line Subpopulation
Description: The criteria for CR, CRi, PR, and nPR are identified in previous outcome measure(s). PD was defined by at least one of the following: the presence of lymphadenopathy; an increase in the previously noted enlargement of the liver or spleen by >/= 50% or the de novo appearance of hepatomegaly or splenomegaly; an increase in the number of blood lymphocytes by >/= 50% with >/= 5000 B-cells per microliter (B-cells/mcL); transformation to a more aggressive histology; or occurrence of cytopenia attributable to CLL. Participants not achieving a CR or PR, and who did not exhibit PD, were considered to have stable disease (SD). The percentage of participants achieving each level of response was calculated as the number of participants meeting the above criteria divided by the number of participants analyzed. The rows below are labeled first by the level of response at the end of 6 cycles (C6), then by level of response at the confirmation assessment.
Time Frame: After 6 treatment cycles and at the confirmation of response assessment at least 12 weeks later (up to 36 weeks)
Population: ITT Population (First-Line Subpopulation)
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 121 | 120
percentage of participants
  CR with biopsy (C6), CR (confirmed) | 21.5 | 9.2
  CR with biopsy (C6), CRi (confirmed) | 2.5 | 0
  CR with biopsy (C6), nPR (confirmed) | 1.7 | 6.7
  CR with biopsy (C6), PR (confirmed) | 19.0 | 17.5
  CR with biopsy (C6), SD (confirmed) | 0 | 1.7
  CR with biopsy (C6), PD (confirmed) | 0 | 0
  CR with biopsy (C6), Missing (confirmed) | 0 | 0
  CR without biopsy (C6), CR (confirmed) | 2.5 | 5.8
  CR without biopsy (C6), CRi (confirmed) | 0 | 0
  CR without biopsy (C6), nPR (confirmed) | 0 | 0
  CR without biopsy (C6), PR (confirmed) | 16.5 | 10.0
  CR without biopsy (C6), SD (confirmed) | 0 | 0
  CR without biopsy (C6), PD (confirmed) | 0 | 0
  CR without biopsy (C6), Missing (confirmed) | 0.8 | 0
  PR (C6), CR (confirmed) | 1.7 | 4.2
  PR (C6), CRi (confirmed) | 0 | 0
  PR (C6), nPR (confirmed) | 0 | 0
  PR (C6), PR (confirmed) | 8.3 | 21.7
  PR (C6), SD (confirmed) | 0 | 0
  PR (C6), PD (confirmed) | 0.8 | 2.5
  PR (C6), Missing (confirmed) | 0 | 0
  SD (C6), CR (confirmed) | 0 | 0
  SD (C6), CRi (confirmed) | 0 | 0
  SD (C6), nPR (confirmed) | 0 | 0
  SD (C6), PR (confirmed) | 0 | 0
  SD (C6), SD (confirmed) | 0 | 0.8
  SD (C6), PD (confirmed) | 0 | 0.8
  SD (C6), Missing (confirmed) | 0 | 0
  Missing (C6), CR (confirmed) | 0.8 | 0
  Missing (C6), CRi (confirmed) | 0 | 0
  Missing (C6), nPR (confirmed) | 0 | 0
  Missing (C6), PR (confirmed) | 0 | 0
  Missing (C6), SD (confirmed) | 0 | 0
  Missing (C6), PD (confirmed) | 0 | 0
  Missing (C6), Missing (confirmed) | 24.0 | 19.2

6. Secondary Outcome: Percentage of Participants Experiencing PD or Death in the First-Line Subpopulation
Description: The criteria for PD are identified in previous outcome measure(s). The percentage of participants experiencing PD or death was calculated as the number of participants with event divided by the number of participants analyzed, multiplied by 100.
Time Frame: End of Cycles 3 and 6 (both treatment arms), end of Cycles 7 to 12 (Rituximab + Chlorambucil arm), after an additional 8 weeks as confirmation of response, then every 3 months for 1 year, then every 6 months until study cutoff (up to 4.5 years)
Population: ITT Population (First-Line Subpopulation)
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 121 | 120
percentage of participants | 27.3 | 46.7

7. Secondary Outcome: Progression-Free Survival (PFS) in the First-Line Subpopulation
Description: The criteria for PD are identified in previous outcome measure(s). PFS was defined as the time from the first dose of trial treatment to the first documentation of PD or death, whichever occurred first. PFS was calculated in months as [first event date minus first dose date plus 1] divided by 30.44.
Time Frame: as for outcome 6
Population: ITT Population (First-Line Subpopulation)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 121 | 120
months | 39.6 [34.3 to NA] — Due to insufficient follow-up among participants assigned to Rituximab + Bendamustine in the first-line subpopulation, a confidence interval upper limit was not reached. | 29.9 [22.4 to 34.4]
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; Unstratified analysis; Test type: Superiority or Other; p = 0.003, Log Rank; Hazard Ratio (HR) = 0.525, 95% CI 2-sided [0.341 to 0.809]
Statistical Analysis 2: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; Stratified analysis: by baseline Binet stage; Test type: Superiority or Other; p = 0.003, Log Rank; Hazard Ratio (HR) = 0.523, 95% CI 2-sided [0.339 to 0.806]

8. Secondary Outcome: Percentage of Participants With Tumor Response of CR or CRi Experiencing PD or Death in the First-Line Subpopulation
Description: The criteria for CR, CRi, and PD are identified in previous outcome measure(s). The percentage of participants experiencing PD or death was calculated as the number of participants with event divided by the number of participants analyzed, multiplied by 100.
Time Frame: as for outcome 6
Population: ITT Population (First-Line Subpopulation); only participants with a tumor response of CR or CRi during study treatment or within 4 months after the end of treatment were considered in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 90 | 77
percentage of participants | 17.8 | 33.8

9. Secondary Outcome: Disease-Free Survival (DFS) in the First-Line Subpopulation
Description: The criteria for CR, CRi, and PD are identified in previous outcome measure(s). DFS was defined as the time from the first assessment of CR or CRi to the first documentation of PD or death, whichever occurred first. DFS was calculated in months as [first event date minus first assessment date of CR/CRi plus 1] divided by 30.44.
Time Frame: as for outcome 6
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 90 | 77
months | 36.8 [32.0 to NA] — Data for > 50% of participants were censored, and thus a confidence interval upper limit was not reached. | 32.0 [22.2 to NA] — Data for > 50% of participants were censored, and thus a confidence interval upper limit was not reached.
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; Test type: Superiority or Other; p = 0.029, Log Rank

10. Secondary Outcome: Percentage of Participants Experiencing PD, Documented Intake of New Leukemia Therapy, or Death in the First-Line Subpopulation
Description: The criteria for PD are identified in previous outcome measure(s). The percentage of participants experiencing PD, intake of new (post-trial) leukemia therapy, or death was calculated as the number of participants with event divided by the number of participants analyzed, multiplied by 100.
Time Frame: as for outcome 6
Population: ITT Population (First-Line Subpopulation)
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 121 | 120
percentage of participants | 29.8 | 49.2

11. Secondary Outcome: Event-Free Survival (EFS) in the First-Line Subpopulation
Description: The criteria for PD and SD are identified in previous outcome measure(s). EFS was defined as the time from the first dose of trial treatment to the first documentation of PD, the beginning of new treatment for any hematologic malignancy, or death from any cause. Those with SD were considered event-free. EFS was calculated in months as [first event date minus first dose date plus 1] divided by 30.44.
Time Frame: as for outcome 6
Population: ITT Population (First-Line Subpopulation)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 121 | 120
months | 39.6 [34.3 to NA] — Data for > 50% of participants were censored, and thus a confidence interval upper limit was not reached. | 29.9 [21.9 to 34.4]
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; Test type: Superiority or Other; p = 0.006, Log Rank

12. Secondary Outcome: Percentage of Participants With Documented Intake of New Leukemia Therapy in the First-Line Subpopulation
Description: The percentage of participants with documented intake of new (post-trial) leukemia therapy was calculated as the number of participants with new therapy divided by the number of participants analyzed, multiplied by 100.
Time Frame: During Cycles 1 to 6 (both treatment arms), Cycles 7 to 12 (Rituximab + Chlorambucil arm), after an additional 8 weeks, then every 3 months for 1 year, then every 6 months until study cutoff (up to 4.5 years)
Population: ITT Population (First-Line Subpopulation)
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 121 | 120
percentage of participants | 9.1 | 18.3

13. Secondary Outcome: Time to Next Leukemia Treatment (TNLT) in the First-Line Subpopulation
Description: TNLT was defined as the time from the first dose of trial treatment to the first documentation of any new leukemia treatment. TNLT was calculated in months as [first new treatment date minus first dose date plus 1] divided by 30.44.
Time Frame: as for outcome 12
Population: ITT Population (First-Line Subpopulation)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 121 | 120
months | NA [NA to NA] — Due to the low number of participants who received new leukemia treatment, the median TNLT could not be calculated. Data for > 90% of participants were censored. | NA [NA to NA] — Due to the low number of participants who received new leukemia treatment, the median TNLT could not be calculated. Data for > 80% of participants were censored.
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; Test type: Superiority or Other; p = 0.037, Log Rank

14. Secondary Outcome: Percentage of Participants With Tumor Response of CR, CRi, PR, or nPR Experiencing PD or Death in the First-Line Subpopulation
Description: The criteria for CR, CRi, PR, nPR, and PD are identified in previous outcome measure(s). The percentage of participants experiencing PD or death was calculated as the number of participants with event divided by the number of participants analyzed, multiplied by 100.
Time Frame: as for outcome 6
Population: ITT Population (First-Line Subpopulation); only participants with a tumor response of CR, CRi, PR, or nPR were considered in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 114 | 107
percentage of participants | 24.6 | 43.9

15. Secondary Outcome: Duration of Response in the First-Line Subpopulation
Description: The criteria for CR, CRi, PR, nPR, and PD are identified in previous outcome measure(s). Duration of response was defined as the time from the first assessment of CR, CRi, PR, or nPR to the first documentation of PD or death, whichever occurred first. Duration of response was calculated in months as [first event date minus first assessment date of CR/CRi/PR/nPR plus 1] divided by 30.44.
Time Frame: as for outcome 6
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 114 | 107
months | 36.8 [31.0 to NA] — Data for > 75% of participants were censored, and thus a confidence interval upper limit was not reached. | 27.7 [20.8 to 40.9]
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; Test type: Superiority or Other; p = 0.007, Log Rank

16. Secondary Outcome: Percentage of Participants Experiencing Death in the First-Line Subpopulation
Description: The percentage of participants experiencing death was calculated as the number of participants with event divided by the number of participants analyzed, multiplied by 100.
Time Frame: as for outcome 6
Population: ITT Population (First-Line Subpopulation)
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 121 | 120
percentage of participants | 14.9 | 15.0

17. Secondary Outcome: Overall Survival (OS) in the First-Line Subpopulation
Description: OS was defined as the time from recorded diagnosis to death from any cause. OS was calculated in months as [death date or last-known alive date minus diagnosis date plus 1] divided by 30.44.
Time Frame: as for outcome 6
Population: ITT Population (First-Line Subpopulation)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 121 | 120
months | 43.8 [39.6 to 43.8] | NA [NA to NA] — Due to insufficient follow-up among participants assigned to Rituximab + Chlorambucil in the first-line subpopulation, the median OS could not be calculated.
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; Test type: Superiority or Other; p = 0.986, Log Rank — Unstratified analysis; Hazard Ratio (HR) = 0.994, 95% CI 2-sided [0.517 to 1.911]
Statistical Analysis 2: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; Stratified analysis: by baseline Binet stage; Test type: Superiority or Other; p = 0.939, Log Rank; Hazard Ratio (HR) = 0.975, 95% CI 2-sided [0.505 to 1.880]

18. Secondary Outcome: Percentage of Participants Achieving Molecular Response in the First-Line Subpopulation
Description: Molecular response was defined as negative minimal residual disease (MRD) during study treatment or within 4 months after the end of treatment. Negative MRD was defined as a proportion of malignant B-cells in normal B-cells < 0.0001. The percentage of participants achieving molecular response was calculated as the number of participants with negative MRD divided by the number of participants analyzed.
Time Frame: Up to 4 months after the last treatment cycle (up to 40 weeks)
Population: ITT Population (First-Line Subpopulation); only participants with a tumor response of CR, CRi, PR, or nPR during study treatment or within 4 months after the end of treatment were considered in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 112 | 106
percentage of participants
  Molecular response | 57.1 | 16.0
  No molecular response | 42.9 | 84.0
Statistical Analysis 1: Comparison: Rituximab + Bendamustine vs Rituximab + Chlorambucil; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected — Based on two-sided continuity corrected Chi-Square Test

19. Secondary Outcome: Number of Participants With Positive and Negative Outcome for MRD in the First-Line Subpopulation
Description: Negative MRD was defined as a proportion of malignant B-cells in normal B-cells < 0.0001, and positive MRD was defined as a proportion of malignant B-cells in normal B-cells >/= 0.0001.
Time Frame: After 6 treatment cycles (up to 24 weeks)
Population: ITT Population (First-Line Subpopulation); only participants with available MRD data (MRD-evaluable participants) were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 78 | 78
participants
  Positive outcome | 30 | 64
  Negative outcome | 48 | 14

20. Secondary Outcome: Proportion of Malignant B-cells in Normal B-cells Among Participants With a Positive Outcome for MRD in the First-Line Subpopulation
Description: The proportion of malignant B-cells in normal B-cells was quantitatively determined, and was calculated as the number of malignant B-cells divided by the number of normal B-cells observed.
Time Frame: After 6 treatment cycles (up to 24 weeks)
Population: ITT Population (First-Line Subpopulation); only participants with a positive outcome for MRD were included in the analysis.
Measure: Mean (Standard Deviation); unit: proportion
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Number analyzed (Participants) | 30 | 64
proportion | 0.0836 (0.22739) | 0.1125 (0.27662)

ADVERSE EVENTS:
Time Frame: From Baseline up to 8 weeks after the start of the last treatment cycle (nonserious adverse events [AEs]; up to 56 weeks) or until the EOT visit (serious AEs; up to 4.5 years)
Description: Based upon the pooled population including both first-line and second line participants
Arm/Group | Rituximab + Bendamustine | Rituximab + Chlorambucil
Serious Adverse Events (participants affected / at risk) | 73/177 | 56/178
Other Adverse Events (participants affected / at risk) | 165/177 | 159/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Bendamustine (N=177) | Rituximab + Chlorambucil (N=178)
Pneumonia (Infections and infestations) | 8 | 2
Herpes zoster (Infections and infestations) | 5 | 0
Lower respiratory tract infection (Infections and infestations) | 4 | 2
Bronchitis (Infections and infestations) | 3 | 2
Neutropenic sepsis (Infections and infestations) | 3 | 3
Infection (Infections and infestations) | 2 | 1
Anal abscess (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Listeria sepsis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Chronic sinusitis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 7
Neutropenia (Blood and lymphatic system disorders) | 6 | 3
Pancytopenia (Blood and lymphatic system disorders) | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac fibrillation (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Pyrexia (General disorders) | 5 | 1
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Ill-defined disorder (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 4
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Blood creatine increased (Investigations) | 1 | 0
International normalized ratio increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adjustment disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Vascular occlusion (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Bendamustine (N=177) | Rituximab + Chlorambucil (N=178)
Neutropenia (Blood and lymphatic system disorders) | 97 | 86
Leukopenia (Blood and lymphatic system disorders) | 42 | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 35 | 41
Anaemia (Blood and lymphatic system disorders) | 40 | 27
Lymphopenia (Blood and lymphatic system disorders) | 30 | 21
Nausea (Gastrointestinal disorders) | 53 | 46
Diarrhoea (Gastrointestinal disorders) | 29 | 20
Constipation (Gastrointestinal disorders) | 27 | 22
Vomiting (Gastrointestinal disorders) | 18 | 20
Abdominal pain (Gastrointestinal disorders) | 3 | 11
Asthenia (General disorders) | 29 | 34
Pyrexia (General disorders) | 33 | 16
Fatigue (General disorders) | 17 | 18
Chills (General disorders) | 16 | 15
Oedema peripheral (General disorders) | 9 | 10
Rash (Skin and subcutaneous tissue disorders) | 28 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Neutrophil count decreased (Investigations) | 8 | 11
Weight decreased (Investigations) | 13 | 5
Headache (Nervous system disorders) | 10 | 14
Dizziness (Nervous system disorders) | 7 | 12
Nasopharyngitis (Infections and infestations) | 10 | 9
Bronchitis (Infections and infestations) | 8 | 9
Infusion related reaction (Injury, poisoning and procedural complications) | 12 | 18
Decreased appetite (Metabolism and nutrition disorders) | 14 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 12
Hypotension (Vascular disorders) | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.